CLINICAL TRIAL: NCT02572739
Title: Assessment of Reliability of Cardiac Output Measurement Based on Impedance (NICCOMO) - Method of Noninvasive Cardiac Output Measurement, Compared to Transthoracic Thermodilution (PiCCO) at Different PEEP Levels
Brief Title: Cardiac Output Measurement With NICCOMO and PiCCO Devices at Different PEEP Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Magdalena Wujtewicz, assistant professor, Medical University of Gdansk
Other Study IDs: GUMed-Wu-002
Record Dates: First submitted 2015-09-23; First posted 2015-10-09 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Diagnostic Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- haemodynamics measuring: those with already implemented PICCO device get impedance device (NICCOMO) attached
  Interventions: Device: PICCO; Device: NICCOMO

INTERVENTIONS:
Device: PICCO — measurements based on thermodilution
Device: NICCOMO — measurements based on impedance

SUMMARY:
Thermodilution cardiac output measurement is a reliable method, but it is an invasive one. PiCCO device requires cannulation of central vein and peripheral artery. Impedance method requires only attachment of special electrodes. Non-invasive methods are less accurate. Aim of study is to assess accuracy and reliability of impedance method ( using NICCOMO device) in comparison of thermodilution method ( using PiCCO device) at different PEEP levels.

DETAILED DESCRIPTION:
Echocardiography is performed prior to measurement to exclude patients with heart valve abnormalities.

Patients without spontaneous ventilation ( deeply unconscious, sedated or sedated and paralysed), ventilated with controlled mechanical ventilation mode with tidal volume 6-8 ml/ideal body weight, resulting in EtCO2 35-45 mmHg, with PiCCO catheters implemented have additionally NICCOMO device attached. Fraction of inspired oxygen (FiO2) is set to achieve saturation >96% at positive end expiratory pressure (PEEP) 0 cmH2O.

Measurement of cardiac output are performed on expiration at PEEP 0, 5, 10, 15 20 cmH2O and at optimal PEEP (obtained from P-V curve). Simultaneously CO value from impedance device is noted. Other haemodynamic parameters, calculated by both devices are also noted - stroke volume (SV), stroke volume variation (SVV), Cardiac index (CI), systemic vascular resistance (SVR), systemic vascular resistance index (SVRI).

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* patients on mechanical ventilation
* circulatory insufficiency (present or in the past) monitored with with PiCCO device

Exclusion Criteria:

* morbid obesity,
* short neck,
* severe pneumonia,
* inability to NICCOMO electrodes attachment,
* massive tissue oedema,
* non-sinus cardiac rhythm,
* tachycardia,
* low cardiac output,
* septic shock,
* heart valve pathologies,
* severe atherosclerosis,
* aortic prosthesis,
* severe hypertension,
* extremes of height and weight,
* intraaortic pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated in intensive therapy unit, mechanically ventilated, haemodynamics monitored with PiCCO technique
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Numbers of measurements of haemodynamic parameters (CO, CI, SV, SVV, CI, SVR, SVRI) obtained with impedance, that differ from those obtained with thermodilution | up to 90 minutes
  measurements taken with impedance and thermodilution simultaneously, at PEEP 0, 5, 10, 15, 20 and at optimal PEEP

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Wujtewicz, Principal Investigator — Department of Ophthalmology, Medical University of Gdańsk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland